CLINICAL TRIAL: NCT06581432
Title: Beamion PANTUMOR-1: A Phase II, Multicentre, Multicohort, Open-label Trial to Evaluate the Efficacy and Safety of Oral Zongertinib (BI 1810631) for the Treatment of Selected HER2-mutated or Overexpressed/Amplified Solid Tumours
Brief Title: Beamion PANTUMOR-1: A Study to Test Whether Zongertinib Helps People With Advanced Cancers With HER2 Alterations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0009; 2023-510429-14-00 (Registry Identifier: CTIS); U1111-1302-3333 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zongertinib treatment (Experimental)
  Interventions: Drug: Zongertinib

INTERVENTIONS:
Drug: Zongertinib — Zongertinib
  Other Names: BI 1810631, Hernexeos®

SUMMARY:
This is a study for people with advanced cancer for whom previous treatment was not successful. Adults aged 18 and over with advanced cancer with HER2 alterations can join the study. The purpose of this study is to find out whether a medicine called zongertinib helps people with advanced cancers with HER2 alterations. HER2 alterations can cause cancer. Zongertinib inhibits HER2.

Participants are put into 13 groups based on the type of advanced cancer and the type of HER2 alterations they have. All participants take one dose of zongertinib each day. Participants can continue the treatment as long as they benefit from it and can tolerate it.

Participants visit the study site regularly. During many of the visits, the doctors check the size of the tumour and whether it has spread to other parts of the body. During all the visits, the doctors check participants' health and take note of any unwanted effects.

ELIGIBILITY:
inclusion criteria:

* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Patients ≥18 years old or over the legal age of consent in countries where that is greater than 18 years at the time of signature of the Informed consent form (ICF).
* Documented (previously established by local testing) Human epidermal growth factor receptor 2 (HER2) status of:

  * HER2 overexpression/amplification
  * Known activating HER2 mutations
* Availability and willingness to provide a sample of archival formalin-fixed paraffin embedded (FFPE) tumour tissue material
* Patient with histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumour who has had at least one prior line of therapy for metastatic disease. In the opinion of the Investigator, patients must be unlikely to tolerate or derive clinically meaningful benefit from further standard of care therapy known to prolong survival.

Further inclusion criteria apply.

exclusion criteria:

* Diagnosis of HER2 mutant Non-small cell lung cancer (NSCLC) (except where there is co-existing presence of HER2 overexpression / amplification)
* Previous or concomitant malignancies other than the 1 treated in this trial within the previous 3 years except:

  * effectively treated non-melanoma skin cancers
  * effectively treated carcinoma in situ of the cervix
  * effectively treated ductal carcinoma in situ of the breast
  * localised prostate cancer on watchful waiting or active surveillance
  * other effectively treated malignancy that is considered cured by local treatment.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Not completely recovered from major surgery (major according to the investigator's assessment) performed prior to screening or planned within 6 months after screening, e.g. hip replacement Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with objective response (OR) | Up to 51 months
  Objective response (OR) is defined as the best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, as assessed by central independent review, from the date of treatment start until the earliest date of progressive disease (PD), death, or last evaluable tumour assessment before the start of subsequent anti-cancer therapy, or trial treatment discontinuation.

SECONDARY OUTCOMES:
Duration of objective response (DOR) | Up to 51 months
  Duration of objective response (DOR) is defined as the time from first documented Objective response (OR) according to RECIST 1.1 until the earliest date of disease progression or death among patients with confirmed OR, assessed by central independent review.
Progression-Free Survival (PFS) | Up to 51 months
  PFS is defined as the time from treatment start until the earliest date of tumour progression according to RECIST 1.1 assessed by central independent review, or death from any cause, whichever occurs first.
Disease control (DC) | Up to 51 months
  Disease control (DC) is defined as best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) where BOR is defined according to RECIST 1.1 from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before the start of subsequent anti-cancer therapy, or treatment discontinuation, as assessed by central independent review.
Occurrence of treatment-emergent Adverse Events (AEs) | Up to 51 months
Change from baseline to Week 48 or progressive disease (PD) by central independent review, if earlier, in the European Organisation for Research and Treatment of Cancer, quality-of-life questionnaire (EORTC QLQ-C30) | At baseline and up to 48 weeks
  QLQ-C30 incorporates both multi-items scales and single-item measures. These include 1 global health status/QoL scale, 5 functional scales, 3 symptoms scales and 6 single items to assess dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. EORTC QLQ-C30 does not produce a single overall summary score by default. Scores can be reported via domain-specific scores or summary score (since 2016) ranging from 0 to 100 with higher scores representing a better QoL.
Overall survival (OS) | Up to 51 months
  OR is defined as the time from start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (80):
- United States (18):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - University of Arizona Comprehensive Cancer Center, Tucson, Arizona
  - Precision NextGen Oncology, Beverly Hills, California
  - Scripps Cancer Center Torrey Pines, La Jolla, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - BRCR Global, Tamarac, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Community MD Anderson Cancer Center - East Medical Oncology, Indianapolis, Indiana
  - Maryland Oncology Hematology, Columbia, Columbia, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Taylor Cancer Research Center, Maumee, Ohio
  - Alliance Cancer Specialists, PC, Wynnewood, Wynnewood, Pennsylvania
  - Sarah Cannon Research Institute at Mary Crowley, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (5):
  - Macquarie University, Macquarie Park, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - Cancer Research South Australia, Adelaide
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
- Canada (5):
  - Cross Cancer Institute (University of Alberta), Edmonton, Alberta
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
- China (8):
  - Peking University First Hospital, Beijing
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Shanghai East Hospital, Shanghai
  - Shanghai GoBroad Cancer Hospital, Shanghai
  - Wuhan Union Hospital, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (6):
  - INS Bergonie, Bordeaux
  - CTR Georges-François Leclerc, Dijon
  - CTR Leon Berard, Lyon
  - HOP Timone, Marseille
  - HOP la Milétrie, Poitiers
  - INS Gustave Roussy, Villejuif
- Germany (5):
  - Justus-Liebig Universität Gießen, Giessen
  - Asklepios Kliniken GmbH & Co. KGaA, Hamburg
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München
- Italy (4):
  - Az. Ospedaliere Umberto I di Ancona, Ancona
  - Istituto Scientifico Romagnolo, Meldola (FC)
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
- Japan (9):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Okayama University Hospital, Okayama, Okayama
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen
- Oslo Universitetssykehus HF, Radiumhospitalet, Oslo, Norway
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Virgen del Rocío, Seville
- United Kingdom (2):
  - Ninewells Hospital & Medical School, Dundee
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link hhttps://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency